CLINICAL TRIAL: NCT04034238
Title: A Phase I Study of Mesothelin-Targeted Immunotoxin LMB-100 in Combination With Tofacitinib in Persons With Previously Treated Pancreatic Adenocarcinoma, Cholangiocarcinoma and Other Mesothelin Expressing Solid Tumors
Brief Title: Mesothelin-Targeted Immunotoxin LMB-100 in Combination With Tofacitinib in Persons With Previously Treated Pancreatic Adenocarcinoma, Cholangiocarcinoma and Other Mesothelin Expressing Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christine Alewine, M.D., Principla Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190128; 19-C-0128
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms With Mesothelin Expression; Epithelioid Mesothelioma; Cholangiocarcinoma, Extrahepatic; Adenocarcinoma, Pancreatic
Keywords: Advanced Cancer; Immunotoxin; Antibody Based Therapeutics; Mesothelin
MeSH Terms: conditions — Cholangiocarcinoma; Adenocarcinoma | interventions — LMB-100; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 1. Dose escalation (Experimental): LMB-100 at escalating doses plus tofacitinib
  Interventions: Drug: LMB-100; Drug: Tofacitinib; Device: Mesothelin Expression
- 2. Dose expansion (Experimental): LMB-100 at optimal dose plus tofacitinib
  Interventions: Drug: LMB-100; Drug: Tofacitinib

INTERVENTIONS:
Drug: LMB-100 — Arms 1 and 2: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
Drug: Tofacitinib — Arms 1 and 2: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
  Other Names: Xeljanz
Device: Mesothelin Expression — Test for mesothelin expression in tumor tissues for study eligibility
  Arms: 1. Dose escalation

SUMMARY:
Background:

The protein mesothelin is found on many kinds of tumors. The drug LMB-100 targets cancer cells that make this protein. Researchers want to see if LMB-100 combined with another drug can help people with these tumors.

Objective:

To find a safe dose of LMB-100 plus tofacitinib in people with pancreatic cancer, bile-duct cancer, and other solid tumors that make mesothelin.

Eligibility:

People ages 18 and older with pancreatic cancer, bile-duct cancer, or any other solid tumor with mesothelin that worsened after treatment or they could not receive standard treatment

Design:

Participants will be screened with:

* Medical history
* Tumor tissue sample. If they do not have a sample, they will have a biopsy.
* Physical exam
* Blood and heart tests
* Scans and x-rays: They may have a dye injected for the scans.

Participants will take the drugs in up to three 21-day cycles. They will take tofacitinib by mouth twice a day on days 1-10 of each cycle. They will have LMB-100 injected into the blood on days 4, 6, and 8 of every cycle. Patients that do not have a medi-port may need to have a central vein access line placed.

Participants will take other drugs on the days they receive LMB-100.

Participants will repeat screening tests during the study. They may have a biopsy at the start of the first 2 cycles.

If participants must stop the study, they will have a safety visit 3-6 weeks after their last dose of the study drug. Some participants may then have visits every 6 weeks.

After treatment, participants will be contacted about once a year. They will be asked about their cancer.

DETAILED DESCRIPTION:
Background:

* Pancreatic cancer is the fourth most common cause of cancer death in the United States, claiming more than 40,000 lives each year.
* Incidence nearly equals mortality with just 6% of participants living five years beyond their diagnosis. Most patients are diagnosed at an advanced stage, but even patients with early-stage disease have a long-term survival of less than 20%.
* Cholangiocarcinoma is a rare disease and just 3,000 patients are diagnosed with the extrahepatic form yearly. The median overall survival of patients with advanced disease receiving standard of care treatment is less than 1 year.
* Expression of mesothelin (MSLN) in pancreatic ductal adenocarcinoma (PDA) has been examined in several published studies and ranges from 86 to 100%. Similar incidence of expression has been observed in extrahepatic cholangiocarcinoma.
* In addition to pancreatobiliary tumors, many other solid tumor types also express MSLN such as mesothelioma, colorectal, lung adenocarcinomas, epithelial ovarian, gastric and triple negative breast cancers, as well as some tumors of squamous cell origin.
* LMB-100 and a closely related immunotoxin also targeting MSLN have been studied in previous Phase 1 clinical studies for mesothelioma and pancreatic cancer.
* Results from these studies showed that almost all patients formed anti-drug-antibodies (ADAs) that neutralized subsequent injection of the product making it ineffective.
* Tofacitinib is an oral Janus Kinase-1 and -3 (JAK) inhibitor approved by the FDA for the treatment of rheumatoid arthritis and ulcerative colitis.
* Pre-clinical studies have shown that tofacitinib can prevent the formation of ADAs against an immunotoxin closely related to LMB-100
* Co-administration of tofacitinib with immunotoxin increased immunotoxin serum half- life in mice and enhanced anti-tumor efficacy
* This clinical trial will investigate whether co-administration of tofacitinib with LMB- 100 can prevent or delay the formation of ADAs and thus allow patients to receive additional effective cycles of LMB-100.

Objectives:

* The primary objective of the dose escalation phase of this study is to assess the safety and tolerability of LMB-100 given in combination with tofacitinib to patients with pancreatic adenocarcinoma, extrahepatic cholangiocarcinoma and other mesothelin-positive solid tumors
* The primary objective of the expansion phase of this study is to determine whether co-administration of tofacitinib delays formation of neutralizing anti-LMB-100 ADAs through cycle 2 of treatment (as measured by LMB-100 serum drug levels) in patients with pancreatobiliary cancers.

Eligibility:

* Age >= 18 years
* Histologically confirmed solid tumor malignancy for which no curative therapy exists
* Participants must have received at least one prior systemic treatment regimen for their disease OR be ineligible to receive available standard treatments for their disease OR refused first-line standard systemic treatments but have been treated with other anti-cancer agents.

Design:

* This is a Phase I study which will accrue up to 45 subjects total, accounting for screen failure.
* Participants will be co-treated for 3 cycles with tofacitinib given orally for the first 10 days of each 21-day cycle, and LMB-100 given on days 4, 6 and 8.
* A 3+3 dose escalation schema will be used. Two dose levels are planned. One minus dose level could be utilized if dose de-escalation is necessary.
* Following identification of an optimal dose and schedule, an expansion phase of 15 participants will be initiated at the optimal dose for patients with pancreatic adenocarcinoma and extrahepatic cholangiocarcinoma. At least 8 participants in the expansion phase must have pancreatic adenocarcinoma.
* Participants on the Dose Escalation and Dose Expansion Arms who appear to be obtaining clinical benefit from LMB-100/tofacitinib after 3 cycles of treatment may elect to receive additional cycles of therapy at the discretion of the principal investigator (PI).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumor malignancy for which no curative therapy exists.
* Pancreatic adenocarcinoma, extrahepatic cholangiocarcinoma or epithelioid subtype of mesothelioma, as determined by National Cancer Institute (NCI) Laboratory of Pathology, OR for all other tumor types, at least 20% of tumor cells must express mesothelin. Determination can be made using archival tumor tissue or fresh biopsy if archival tumor tissue is not available.
* All patients must have evaluable disease (i.e., measurable per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. or by following carbohydrate antigen 19-9 (CA19-9) tumor marker). Patients in the expansion cohort must have measurable disease, per RECIST 1.1. evaluation of measurable disease.
* Patients must have received at least one prior standard systemic treatment regimen for advanced disease OR be ineligible to receive available standards due to co-morbidities, prior toxicity, lack of standard options for tumor type, or having received all standards available for prior treatment of early-stage disease OR have refused first-line standard systemic treatment but have received prior anti-cancer treatments.
* Patients with deficient Mismatch Repair (dMMR)/high levels of MicroSatellite Instability (MSI-H) disease must have received at least one prior anti-programmed cell death 1 (PD1) therapy, be ineligible to receive this treatment due to concurrent medical conditions or have refused this therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of LMB-100 alone or in combination with tofacitinib in persons with <18 years of age, children are excluded from this study.
* Patients must be more than 14 days removed from most recent minor surgical procedure (such as biliary stenting), 28 days from most recent major surgical procedure and 14 days from radiation therapy, systemic treatments (such as chemotherapy), or experimental drug treatment. All acute toxicities from prior treatment must have resolved to grade 1 or less except alopecia, anemia, peripheral neuropathy, or endocrinopathies corrected by replacement therapy.
* Adequate hematological function: neutrophil count of >= 1.5 x 10^3 cells/micro liters, platelet count of >= 85,000/micro liters, hemoglobin greater than or equal to 9 g/dL
* Serum albumin >= 2.5 mg/dL without intravenous supplementation
* Adequate liver function: Bilirubin <2.5 x upper limit of normal (ULN) for all, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN except for patients with significant tumor burden in their liver where AST and ALT < 5x ULN is acceptable in the absence of other etiologies for transaminitis
* Adequate renal function: creatinine clearance [Estimating glomerular filtration rate (EGFR) method or measured] >= 50 mL/min. Measured clearance will be used if both numbers are available.
* Must have left ventricular ejection fraction >= 50%
* Must have an ambulatory oxygen saturation of > 88% on room air
* The expansion phase patients must meet all eligibility criteria above AND must have diagnosis of pancreatic adenocarcinoma or extrahepatic cholangiocarcinoma with pathology confirmed to be consistent with one of these diagnoses by NCI Laboratory of Pathology.
* The effects of LMB-100 alone or in combination with tofacitinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry until 3 months the last dose of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases as CNS penetration of LMB-100 is expected to be poor. CNS metastases are permitted if they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days.
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant pulmonary disease other than that related to the primary cancer, uncontrolled diabetes mellitus, and/or significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina, or clinically significant pericardial effusion).
* Any known diagnoses, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition (other than mesothelin [+] cancer diagnosis) that would contraindicate the use of an investigational drug, interfere with tumor measurement or lead to a life expectancy of less than 6 months as judged by the investigator.
* Contraindication to receiving prophylactic doses of low-molecular weight heparin (LMWH) or direct oral anticoagulants (DOAC) such as current active bleeding (except for grade 1 hematuria or epistaxis), recent history of significant bleeding without subsequent effective medical or surgical intervention, known history of gastric varices, uncontrolled malignant hypertension, history of coagulopathy that confers increased risk of bleeding. Patients on concurrent treatment with anti-platelet agents such as aspirin or clopidogrel are eligible if deemed to have acceptable risk of bleeding in consultation with Hematologist. Patients already receiving prophylactic or therapeutic doses of anticoagulant (heparin-based, or DOAC) for at least 4 weeks with no indication of significant bleeding while on therapy are considered NOT to have a contraindication to this therapy.
* Inability to administer or unwillingness to comply with recommended venous thromboembolism (VTE) prophylaxis for the duration of study treatment.
* Prior diagnosis of hematologic malignancy
* Active or uncontrolled infections (including tuberculosis, human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) or reasonable clinical suspicion of an active infection (such as cholangitis) as tofacitinib suppresses lymphocyte signaling and will impair host response to infection
* Latent tuberculosis (TB) infection as identified by interferon-gamma release assay (IGRA). If IGRA is indeterminate, tuberculin skin test (TST) may be used to determine status.
* Live attenuated vaccinations within 14 days prior to treatment.
* Use of a strong inhibitor or inducer of cytochrome P450 3A4 (CYP3A4) within 14 days prior to enrollment or similarly updated source for a list of such agents)
* Inability to take or digest oral medication.
* Dementia or altered mental status that would prohibit informed consent.
* Pregnant women are excluded from this study because the effects of LMB-100 and/or tofacitinib on the developing fetus are unknown and may have the potential to cause teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100 and/or tofacitinib, breastfeeding should be discontinued if the mother is treated with either of these agents.
* Baseline corrected QT interval by Fredericia (QTcF) interval of > 470 ms, participants with baseline resting bradycardia < 45 beats per minute, or baseline resting tachycardia >100 beats per minute.
* Participants with contra-indication and/or history of severe hypersensitivity reactions to any components related to LMB-100 and tofacitinib.
* Patients who have previously received LMB-100 (and therefore have high-levels of preexisting anti-drug antibodies (ADAs) to drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Alewine, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Skorupan N, Peer CJ, Zhang X, Choo-Wosoba H, Ahmad MI, Lee MJ, Rastogi S, Sato N, Yu Y, Pegna GJ, Steinberg SM, Kalsi SS, Cao L, Figg WD, Trepel JB, Pastan I, FitzGerald D, Alewine C. Tofacitinib to prevent anti-drug antibody formation against LMB-100 immunotoxin in patients with advanced mesothelin-expressing cancers. Front Oncol. 2024 Apr 19;14:1386190. doi: 10.3389/fonc.2024.1386190. eCollection 2024. PMID 38706610
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0128.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3/19 subjects were enrolled but not treated (2 in Dose Escalation phase, and 1 in Dose Expansion phase). No data were collected for these participants.
Groups:
- Dose Escalation- Dose Level 1 LMB-100 100 mcg/kg: LMB-100 at escalating doses plus tofacitinib
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
  Mesothelin Expression: Test for mesothelin expression in tumor tissues for study eligibility
- Dose Escalation- Dose Level 2 - LMB -100 140 mcg/kg: LMB-100 at escalating doses plus tofacitinib
  LMB-100: Arms 2: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 2: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
  Mesothelin Expression: Test for mesothelin expression in tumor tissues for study eligibility
- Dose Expansion LMB-100 100 mcg/kg: LMB-100 at optimal dose plus tofacitinib
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
- Enrolled But Not Treated: Participants were enrolled but not treated.
Period: Dose Escalation Phase
Arm/Group | Dose Escalation- Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation- Dose Level 2 - LMB -100 140 mcg/kg | Dose Expansion LMB-100 100 mcg/kg | Enrolled But Not Treated
Started | 7 | 3 | 0 | 2
Completed | 6 | 3 | 0 | 0
Not Completed | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Screen failures | 0 | 0 | 0 | 2
Period: Dose Expansion Phase
Arm/Group | Dose Escalation- Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation- Dose Level 2 - LMB -100 140 mcg/kg | Dose Expansion LMB-100 100 mcg/kg | Enrolled But Not Treated
Started | 0 | 0 | 6 | 1
Completed | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 1 | 1
Not completed — Not treated due to study hold. | 0 | 0 | 0 | 1
Not completed — Discontinued treatment before received LMB-100 during first cycle | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Dose Level 1 LMB-100 100 mcg/kg: LMB-100 at escalating doses plus tofacitinib
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
  Mesothelin Expression: Test for mesothelin expression in tumor tissues for study eligibility
- Dose Escalation Dose Level 2 LMB-100 140 mcg/kg: LMB-100 at escalating doses plus tofacitinib
  LMB-100: Arms 2: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 2: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
  Mesothelin Expression: Test for mesothelin expression in tumor tissues for study eligibility
- Dose Expansion LMB-100, 100 mcg/kg: LMB-100 at optimal dose plus tofacitinib
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg | Total
Number analyzed (Participants) | 7 | 3 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 2 | 9
  >=65 years | 2 | 1 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.79 (15.99) | 54.53 (16.26) | 70.68 (11.36) | 63.76 (14.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 5
  Male | 3 | 2 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 2 | 7
  Unknown or Not Reported | 3 | 1 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 6 | 3 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of LMB-100 With Tofacitinib
Description: MTD is defined as the maximum dose at which less than 33% of participants experience a dose-limiting toxicity (defined as any events occurring within the first cycle of treatment (21 days) such as any death not clearly due to the underlying disease or extraneous causes).
Time Frame: First cycle of treatment (21 days)
Measure: Number; unit: mcg/kg given days 4, 6, 8 every cycle
Groups:
- All Participants in Dose Escalation Dose Level 1, and Dose Level 2: All Participants in Dose Escalation Dose Level 1, and Dose Level 2 administered LMB-100: Both Arms intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 and Tofacitinib orally twice daily on days 1-10 of each cycle, and LMB-100.
Arm/Group | All Participants in Dose Escalation Dose Level 1, and Dose Level 2
Number analyzed (Participants) | 10
mcg/kg given days 4, 6, 8 every cycle | 100

2. Primary Outcome: Percentage of Participants With Pancreatobiliary Cancer and LMB-100 Plasma Drug Levels Above Threshold 600ng/mL During Cycle 2 Who Received LMB-100 at Maximum Tolerated Dose
Description: This measure assessed how many participants have LMB-100 plasma drug levels higher than threshold (600 ng/mL) during Cycle 2 pharmacokinetics (PK) measurements, a sign of effective prevention of anti-LMB-100 antibodies. The validated enzyme-linked immunosorbent assay (ELISA) test was used to measure plasma LMB-100 concentration. Below 600ng/mL is considered a bad outcome and above 600ng/mL is considered a good outcome.
Time Frame: Plasma LMB-100 levels during Cycle 2 treatment (each cycle = 21 days)
Population: Per protocol, this measure includes all participants who meet eligibility criteria for the dose expansion (pancreatobiliary diagnosis) and received LMB-100 at the Maximum Tolerated Dose (Dose Escalation-Dose Level 1 (DL1) and Dose expansion, n =11). Only participants who have pharmacokinetics results during Cycle 2 are evaluable. Five more participants were not evaluable due to not receiving Cycle 2 treatment or not having pharmacokinetics results.
Measure: Number; unit: Percentage of participants
Groups:
- Dose Expansion LMB-100, 100 mcg/kg: LMB-100 at optimal dose plus tofacitinib - 100 mcg/kg LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
Arm/Group | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 6
Percentage of participants | 33.3

3. Primary Outcome: Number of Participants With Serious Adverse Events Possibly, Probably, and/or Definitely Related to LMB-100 Treated in the Dose Escalation Group
Description: Grade 1-5 adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 observed in participants with pancreatic cancer. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant. Grade 4 is life-threatening consequences. Grade 5 is death related to adverse events.
Time Frame: Throughout study treatment until 30 days post-completion, approximately 13 weeks
Population: Per protocol, this outcome measure was only assessed in the dose escalation dose level 1 and dose escalation dose level 2 groups.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Dose Level 1 LMB-100 100 mcg/kg: LMB-100 100 mcg/kg
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
- Dose Escalation Dose Level 2 LMB-100 140 mcg/kg: LMB-100 140 mcg/kg
  LMB-100: Arms 2: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 2: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg
Number analyzed (Participants) | 7 | 3
Participants | 1 | 2

4. Secondary Outcome: Percentage of Participants With LMB-100 Plasma Drug Levels Above Threshold 600ng/mL During Cycle 2 in Dose Escalation
Description: This measure assessed how many participants in the dose escalation have LMB-100 plasma drug levels higher than threshold (600 ng/mL) during Cycle 2 pharmacokinetics (PK) measurements, a sign of effective prevention of anti-LMB-100 antibodies. The validated enzyme-linked immunosorbent assay (ELISA) test was used to measure plasma LMB-100 concentration. Below 600ng/mL is considered a bad outcome and above 600ng/mL is considered a good outcome.
Time Frame: Plasma LMB-100 levels during Cycle 2 of treatment (each cycle = 21 days)
Population: 6/10 participants were not evaluable for this endpoint because they did not receive the second cycle of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg
Number analyzed (Participants) | 4 | 0
Percentage of participants | 75 |

5. Secondary Outcome: Maximum Observed (Peak) Plasma Concentration (Cmax) of LMB-100
Description: The maximum observed analyte concentration in plasma was reported.
Time Frame: Pre-administration, end-of-infusion, then 1, 2, 4, 8-10, 12-16 hours post- LMB-100 during cycle 1 (each cycle = 21 days)
Population: 1/6 participants from the expansion cohort were not evaluable because they discontinued treatment before receiving LMB-100 during their 1st cycle.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 7 | 3 | 5
ng/mL | 1644.43 (343.08) | 2160.67 (797.9) | 1466.4 (257.25)

6. Secondary Outcome: Percentage of Participants Without Delayed Formation of Neutralizing Anti-LMB-100 Anti-drug Antibodies (ADAs)
Description: This measure assessed how many participants have no LMB-100 plasma drug levels higher than threshold (600 ng/mL) during Cycle 3 pharmacokinetics (PK) measurements, a sign of effective prevention of anti-LMB-100 antibodies. The validated enzyme-linked immunosorbent assay (ELISA) test was used to measure plasma LMB-100 concentration. Below 600ng/mL is considered a bad outcome and above 600ng/mL is considered a good outcome.
Time Frame: Plasma LMB-100 levels during Cycle 3 treatment (each cycle = 21 days)
Population: 12/16 participants were not evaluable because they did not receive a 3rd cycle of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1
Percentage of participants | 100 | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUC(INF)) of LMB-100
Description: AUC is a measure of the serum concentration of LMB-100 over time. It is used to characterize drug absorption.
Time Frame: as for outcome 5
Population: 3/16 participants from both cohorts were not analyzed they did not have AUC(INF) of LMB-100 measured during the 1st cycle (i.e., Not evaluable)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 6 | 2 | 5
h*ng/mL | 2415.9 (1041.2) | 2918.5 (2434.6) | 2804.1 (190.14)

8. Secondary Outcome: Plasma Half-Life (T1/2) of LMB-100
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 5
Population: 3/16 participants were not analyzed because they did not have Plasma Half-life (T1/2) of LMB-100 measured during the 1st cycle (i.e., Not evaluable).
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 6 | 2 | 5
hour (h) | 1.0 (0.39) | 0.8 (0.22) | 1.2 (0.25)

9. Secondary Outcome: Number of Participants With Serious Adverse Events Possibly, Probably, and/or Definitely Related to LMB-100 Who Have Pancreatobiliary Cancer
Description: Grade 1-4 adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 observed in participants with pancreatic cancer. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant. Grade 4 is life-threatening consequences. Grade 5 is death related to adverse event.
Time Frame: Throughout study treatment until 30 days post-completion, approximately 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 6
Participants | 4

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Regardless of Attribution Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Throughout study treatment until 30 days post-completion, approximately 13 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation- Dose Level 1 LMB-100 100 mcg/kg: LMB-100 100 mcg/kg
  LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
Arm/Group | Dose Escalation- Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
Number analyzed (Participants) | 7 | 3 | 6
Participants | 7 | 3 | 6

11. Other Pre Specified Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: A dose limiting toxicity is defined as any events occurring within the first cycle of treatment (21 days) such as any death not clearly due to the underlying disease or extraneous causes, transaminitis that meets criteria for Hy's Law: grade ≥2 elevation of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) with simultaneous elevation of total bilirubin to ≥ 2x ULN while alkaline phosphatase remains < 2x upper limit of normal (ULN). Some hematological toxicities, and Grade ≥3 non-hematological toxicities; and any other drug related toxicity considered significant enough to be qualifies as a DLT in the opinion of the principal investigator. Inability to start cycle 2 within 2 weeks after completing cycle 1 due to drug-related adverse events.
Time Frame: First cycle (21 days)
Population: 1 of 7 participants in Dose Escalation-Dose Level 1 is not evaluable due to withdrawal from the study with loss of follow-up before the conclusion of the DLT period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg
Number analyzed (Participants) | 6 | 3
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Throughout study treatment until 30 days post-completion, approximately 13 weeks.]
Groups:
- Dose Expansion LMB-100, 100 mcg/kg: LMB-100 at optimal dose plus tofacitinib - 100 mcg/kg
  LMB-100 at optimal dose plus tofacitinib LMB-100: Arms 1: Administered intravenous (IV) as an approximate 30-minute infusion of each 21-day cycle on days 4, 6 and 8 until disease progression, intolerance or withdrawal from study.
  Tofacitinib: Arms 1: Administered orally twice daily on days 1-10 of each cycle until disease progression, intolerance or withdrawal from study.
Arm/Group | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg | Dose Expansion LMB-100, 100 mcg/kg
All-Cause Mortality (participants affected / at risk) | 6/7 | 2/3 | 4/6
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/3 | 4/6
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg (N=7) | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg (N=3) | Dose Expansion LMB-100, 100 mcg/kg (N=6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Intraoperative complication (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Dose Level 1 LMB-100 100 mcg/kg (N=7) | Dose Escalation Dose Level 2 LMB-100 140 mcg/kg (N=3) | Dose Expansion LMB-100, 100 mcg/kg (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 2 (4) | 1 (3)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (12) | 2 (2) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 5 (10) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (9) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 1 (1) | 4 (4)
Fever (General disorders) | 1 (4) | 2 (2) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (12) | 3 (3) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (9) | 1 (3) | 4 (9)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (4)
Immune system disorders - Other, Inflammatory Synovitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — laceration of the nasal dorsum from mechanical fall
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Localized edema (General disorders) | 4 (4) | 0 (0) | 2 (4)
Lymphocyte count decreased (Investigations) | 4 (10) | 3 (8) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (4) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other, verruca lesion" (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (6) | 1 (1) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (4) | 1 (1)
White blood cell decreased (Investigations) | 1 (2) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04034238/Prot_SAP_000.pdf
  • Informed Consent Form: Screening Consent (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT04034238/ICF_001.pdf
  • Informed Consent Form: Standard Consent (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT04034238/ICF_002.pdf